CLINICAL TRIAL: NCT03302871
Title: Integrated Management With Brain Stimulation and Hybrid Training Enhances Functional Gains in Children With Cerebral Palsy Treated by Botulinum Toxin A
Brief Title: Integrated Management Enhances Functional Gains in Children With Cerebral Palsy Treated by BoNT-A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Nigar Dursun, Professor, MD, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KOUKAEK 2016/20
Record Dates: First submitted 2017-10-02; First posted 2017-10-05 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; botulinum toxin A; constraint induced movement therapy; transcranial direct current stimulation
MeSH Terms: conditions — Cerebral Palsy | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA; Transcranial Direct Current Stimulation; 2-(4-ethoxybenzyl)-1-diethylaminoethyl-5-isothiocyanatobenzimidazole; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntensive Therapy Group (Experimental): Children who received Botulinum toxin type A to plegic upper limb would be treated by transcranial direct current stimulation and a hybrid training model of CIMT and BIT
  Interventions: Drug: Botulinum toxin type A; Device: transcranial direct current stimulation; Other: hybrid training model of CIMT and BIT
- Control Group (Active Comparator): Children who received Botulinum toxin type A to plegic upper limb would continue their usual care
  Interventions: Drug: Botulinum toxin type A; Other: usual care

INTERVENTIONS:
Drug: Botulinum toxin type A
  Other Names: Botox, Dysport
Device: transcranial direct current stimulation
  Other Names: noninvasiv brain stimulation
  Arms: İntensive Therapy Group
Other: hybrid training model of CIMT and BIT
  Arms: İntensive Therapy Group
Other: usual care
  Other Names: physical therapy
  Arms: Control Group

SUMMARY:
Evidence from literature support the use of Botulinum toxin A (BoNT-A) for upper limb spasticity management in children with cerebral palsy (CP). Constraint Induced Movement Therapy (CIMT) and Bilateral Intensive Training (BIT) are indicated as effective and complimentary treatments to improve motor function in these children. In a recent trial combined noninvasiv brain stimulation and CIMT enhanced therapy induced functional gains.

In this clinical trial the aim was to evaluate the effects of transcranial direct current stimulation (t-DCS) plus intensive hybrid training model of modified CIMT and BIT when integrated with BoNT-A treatment in children with unilateral CP.

DETAILED DESCRIPTION:
Although BoNT-A is effective in spasticity management there is inconclusive evidence to support its usage for improvement in upper limb activity and function. Combination of BoNT-A and occupational therapy (OT) is found to be more effective then OT alone in reducing impairment, improving activity level and goal achievement. Intensive hybrid training models of CIMT and BIT and noninvasive brain stimulation are promising treatments on motor learning in children with CP. The aim of this clinical trial is to show the additional gains that could be provided by an integrated treatment of transcranial direct current stimulation (t-DCS) plus intensive hybrid training model of modified CIMT and BIT to BoNT-A injections in children with unilateral CP.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of unilateral cerebral palsy
* able to activate wrist and finger extensors
* being scheduled for BoNT-A treatment for upper limb

Exclusion Criteria:

* significant loss of wrist and or fingers
* history of orthopedic surgery to plegic upper limb

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2016-01-18 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Assisting Hand Assesment | 6 weeks
  Bilateral Hand Function Evaluation Instrument

SECONDARY OUTCOMES:
Jebsen Taylor Hand Function Test | 6 weeks
  Unilateral Hand Function Evaluation Instrument

OTHER OUTCOMES:
Modifed Ashworth Scale | 6 weeks
  Measurement of Tone
Active ROM of wrist dorsiflexion | 6 weeks
  Measurement of active muscle function
Modified Tardieu Scale | 6 weeks
  Measurement of spasticity

CONTACTS AND LOCATIONS:
Overall Officials: Nigar Dursun, MD, Principal Investigator — Kocaeli University
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No